CLINICAL TRIAL: NCT06924099
Title: Tumor Treating Fields General Routine Clinical Care in Newly Diagnosed Glioblastoma Patients: a French Prospective Non-Interventional Study - TIGER France
Brief Title: TTFields General Routine Clinical Care in ndGBM Patients: a French Prospective Non-Interventional Study (TIGER France)
Acronym: TIGER France
Status: Recruiting | Type: Observational
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TIGER France
Record Dates: First submitted 2024-09-18; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-05

CONDITIONS: Glioblastoma
Keywords: newly diagnosed Glioblastoma (GBM); Tumor Treating Fields - TTFields
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective multicenter non-interventional study (NIS) aims at confirming the survival benefit of Optune Gio® - in terms of OS and PFS - and describing device usage (compliance will be measured through patient's usage report, recorded by each device) and impact on QoL, in a real-life setting in France, in a large cohort of participants with newly diagnosed GBM who completed radiotherapy and concomitant TMZ after surgery and initiatingtreatment with Optune Gio® device together with maintenance TMZ.

A special emphasis will be given to the evaluation of QoL and the impact of Optune Gio® on daily life, considering the limited life expectancy of these patients, the symptom burden and significant disease-related disability.

DETAILED DESCRIPTION:
GBM is one of the most common malignant primary brain tumor in adults with an overall incidence in Europe and in France of approximately 3/100,000. In France, 2,233 patients were estimated to be diagnosed with histologically-confirmed GBM in France in 2020. GBM are particularly aggressive and treatment resistant, with a 5-year overall survival (OS) of only 7.0 % in France. Since 2005, standard treatment for newly diagnosed GBM consists of maximal feasible surgical resection or biopsy followed by standard brain radiation therapy with concomitant temozolomide (TMZ) and a further 6 cycles of TMZ alone (Stupp protocol). This treatment demonstrated a significant increase in median OS compared to surgery and radiotherapy alone (14.6 vs 12.1 months).

Since 2005, despite several of phase III clinical trials conducted, TTFields treatment was the first to report a significant improvement in GBM patients' survival compared to the previous standard of care. This pivotal phase III clinical trial randomized 695 patients with newly diagnosed GBM receiving either TTFields plus maintenance TMZ or TMZ alone, after completion of standard radiochemotherapy. Adding TTFields to maintenance TMZ significantly improved median progression-free survival (PFS) and median OS compared to TMZ alone. Impact of TTFields on survival appeared comparable to that achieved by the addition of TMZ to radiotherapy.

These results led to FDA approval of Optune Gio® and to CE mark in the European Union in association with maintenance TMZ in patients with newly diagnosed GBM, after surgery and radiotherapy with adjuvant TMZ. Optune Gio® obtained national reimbursement in several European countries in this indication, as Germany, Switzerland, Sweden and France. The National Commission for the Evaluation of Medical Devices and Health Technologies (CNEDiMTS) issued on 20 July 2021 a positive opinion to Optune Gio® for inclusion into the reimbursement list in the following indication: "in association with maintenance TMZ, after surgery and radiochemotherapy in patients with newly diagnosed GBM, as part of a shared decision between the patient and the medical team".

This prospective multicenter non-interventional study (NIS) aims at confirming the survival benefit of Optune Gio® - in terms of OS and PFS - and describing device usage (compliance will be measured through patient's usage report, recorded by each device) and impact on QoL, in a real-life setting in France, in a large cohort of participants with newly diagnosed GBM who completed radiotherapy and concomitant TMZ after surgery and initiating treatment with Optune Gio® device together with maintenance TMZ.

A special emphasis will be given to the evaluation of QoL and the impact of Optune Gio® on daily life, considering the limited life expectancy of these patients, the symptom burden and significant disease-related disability.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged ≥ 18 years old.
* Participant with newly diagnosed GBM.
* Participant who completed radiochemotherapy after surgery or biopsy.
* Participant within first 2 cycles of maintenance TMZ.
* Participant for whom the physician has decided to initiate treatment with Optune® according to Instruction For Use or medical guidelines.

Exclusion Criteria:

* Participant currently participating in a prospective clinical trial studying a different treatment than the one studied in this current prospective study.
* Patient currently breastfeeding.
* Patient who is pregnant, thinks she might be pregnant or is trying to become pregnant. Patient of childbearing potential must use a contraceptive method for the whole duration of their participation in the study.
* Patient suffering from a significant neurological disease (primary epilepsy, dementia, progressive degenerative neurological disorder, meningitis or encephalitis, hydrocephalus associated with increased intracranial pressure).
* Patient with a known sensitivity to conductive hydrogels, such as gel used with electrocardiogram (ECG) or transcutaneous electrical nerve stimulation (TENS) electrodes.
* Patient with an active implanted medical device, a cranial defect (such as a missing bone that has not been replaced) or bullet fragments. Active electronic devices include, for example, deep brain stimulators, spinal cord stimulators, vagus nerve stimulators, pacemakers and defibrillators.
* Participant being deprived of liberty by a judicial or administrative decision, or who is under a measure of legal protection (e.g. guardianship or curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tdb
Sampling Method: Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 18 months (mean FU time)
  OS, defined as the time from the date of treatment initiation with Optune® to the date of death from any cause. Participants still alive at the time of the statistical analysis will be censored at the date they were last known to be alive

SECONDARY OUTCOMES:
Health Related Quality of life - European Organization for Research and Treatment of Cancer C30 questionnaire | at start of TTFields treatment, at month 2, month 4, month 6, month 12 and month 18 after start of TTFields treatment
  QoL will be assessed by the EORTC quality-of-life questionnaire. The EORTC QLQ-C30 is a 30-item questionnaire designed to assess the Health-Related Quality ofLife (HRQoL) of cancer patients that has been validated in brain cancer. It incorporates multi-item scales: functional scales (physical, role, cognitive, emotional, and social); symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale. The items on the EORTC QLQ-C30 measures are scaled, scored, and transformed to a linear scale (0 -100) with a higher score representing a higher level of symptoms.
Health Related Quality of life - European Organization for Research and Treatment of Brain Cancer BN20 questionnaire | at start of TTFields treatment, at month 2, month 4, month 6, month 12 and month 18 after start of TTFields treatment
  QoL will be assessed by the EORTC quality-of-life questionnaire. The EORTC QLQ-BN20, specifically developed and validated for patients with brain cancer, includes 20 items assessing visual disorder, motor dysfunction, various disease symptoms, treatment toxicity, and future uncertainty. The items on the EORTC QLQ-BN20 measures are scaled, scored, and transformed to a linear scale (0 -100) with a higher score representing a higher level of symptoms.
Usage of Optune Gio® | at start of TTFields treatment, month 2 and month 4 after start of TTFields treatment
  The 2 device specific questionnaires Optune Gio® initiation and follow-up were developed by Novocure to evaluate the factors influencing participants' decision to initiate treatment with Optune Gio® and the impact of Optune Gio® treatment on participants' daily life. The Optune Gio® initiation questionnaire will be administered before the initiation of Optune Gio® treatment. This questionnaire consists of 9 questions:
  3 questions relate to the information about Optune Gio® received by the participants (when, how long and with whom) 6 questions relate to the factors influencing participants' decision to initiation Optune Gio® treatment: 5 questions answered using a 5-point Likert scale from not at all to very much plus one free text question.
  The Optune Gio® follow-up questionnaire will be administered 2 and 4 months after Optune Gio® treatment initiation. It consists of 6 questions, each of them answered using a 5-level Likert scale from not at all to much more than expected.
Progression Free Survival | through study completion, an average of 18 months (mean follow-up time)
  PFS under TTFields treatment, defined as the time from the date of treatment initiation with Optune® to the date of first documented radiological progression reported by investigators or death from any cause.
Optune Gio® safety profile and deficiencies | through study completion, an average of 18 months (mean follow-up time)
  All non-serious AEs will be assessed according to incidence and causality. All SAEs will be assessed according to incidence, grade, causality, outcome, and action taken. Potential DDs of Optune® device that might have led to a SAE if no action had been taken will also be collected and presented descriptively.

CONTACTS AND LOCATIONS:
Locations (24):
- France (24):
  - Chu Amiens Picardie, Amiens
  - Institut Sainte-Catherine, Avignon
  - Chu Saint Andre, Bordeaux
  - Chu Brest Hopital Morvan, Brest
  - Hopital Neurologie Pierre Wetrheimer, Bron
  - Crlcc Francois Baclesse, Caen
  - Centre Lutte Contre Le Cancer Jean Perrin, Clermont-Ferrand
  - Crlcc Georges Francois Leclerc, Dijon
  - Chu de Grenoble Alpes, La Tronche
  - Hopital Roger Salengro, Lille
  - Centre Hospitalier La Timone, Marseille
  - Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier
  - CHU de Nice, Nice
  - CHU de Nîmes - HOPITAL CAREMEAU, Nîmes
  - Ch Regional Orleans, Orléans
  - Hopital Saint Louis, Paris
  - Gh Pitie Salpetriere Aphp, Paris
  - CRLCC - Centre Eugène Marquis, Rennes
  - Crlcc Henri Becquerel, Rouen
  - Chu de Saint Etienne, Saint-Priest-en-Jarez
  - Hopital Foch, Suresnes
  - Hia Sainte Anne, Toulon
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No